CLINICAL TRIAL: NCT01881334
Title: A Compassionate Release Protocol: Expanded Access to T-cell Depleted Haplo-Identical Stem Cells for Patients Receiving Allogeneic Transplantation Using a Related Haplo-Identical Donor and Unrelated, Umbilical Cord Blood Donor(s) for the Treatment of High Risk Malignancies or Non-Malignant Disorders Requiring Allogeneic Transplantation
Brief Title: Expanded Access to T-cell Depleted Haplo-Identical Stem Cells for Patients Receiving Haplo-Identical and Unrelated Cord Blood Transplants
Status: Available | Type: Expanded Access
Sponsor: Joanne Kurtzberg, MD (Other)
Collaborators: Duke University (Other); Miltenyi Biotec, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, MD, Duke University
Organization: Duke University (Other)
Other Study IDs: Pro00045700
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hematologic Malignancies; Inborn Errors of Metabolism Disorders; Immune Deficiencies
Keywords: Haploidentical Donor; T-cell depleted Stem Cells; Allogeneic Transplant; Umbilical Cord Blood Donor; High Risk Malignancies; Metabolic Disorders; Immune Deficiency; Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia; Myelodysplastic Syndrome; ALL; AML; MDS; CGD; SCID; Adrenoleukodystrophy; Metachromaticleukodystrophy; Krabbe; PMD; Hunter's; Hurler's; Severe Aplastic Anemia; Lymphoma; Sickle Cell Disease; Thalassemia
MeSH Terms: conditions — Hematologic Neoplasms; Metabolic Diseases; Immunologic Deficiency Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Adrenoleukodystrophy; Anemia, Aplastic; Lymphoma; Anemia, Sickle Cell; Thalassemia

INTERVENTIONS:
Biological: CliniMACS CD34 Reagent System — The CliniMACS CD34 Reagent System is a medical device that is used in vitro to select and enrich CD34+ cells from heterogeneous hematologic cell populations for transplantation in cases where this is clinically indicated.

SUMMARY:
The objective of this study is to make T-cell depleted stem cells from a family member who is a half match (haplo-identical) available on an expanded access basis to patients receiving one or two unrelated cord blood transplants who are at a higher risk of not engrafting in a safe amount of time. The purpose of the related stem cells is to give the bone marrow a "jump start" towards recovery. Ultimately, the cord blood cells will grow and permanently rescue the bone marrow.

DETAILED DESCRIPTION:
The primary purpose of the study is to provide expanded access of T-cell depleted haplo-identical stem cells for patients receiving allogeneic transplantation from a related haplo-identical donor and an unrelated, umbilical cord blood (UUCB) unit(s) for the treatment of high risk malignancies and non-malignant disorders. The T-cell depleted haplo-identical stems cells are intended to facilitate early, short-term myeloid engraftment with the primary goal of minimizing early infections and other non-relapse mortality while the UUCB cells engraft as the durable and permanent graft. Patients with high risk or refractory malignancies, or non-malignant disorders amenable to stem cell transplantation therapy but lacking conventional related or unrelated donors will be eligible for this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Have a consenting related haplo-identical (3/6, 4/6, or 5/6 if DRB1 mismatch) stem cell donor.
* Have one or two available 4, 5, or 6/6 antigen matching unrelated UCB unit(s) that will deliver a total cell dose >3.0 x 10e7 cells/kg. Patients who do not have a single UCB unit that will deliver the minimum required cell dose, two partially HLA-matched UCB units which together meet the minimum cell dose requirement, can be used for 1 transplant. These units must be HLA-matched minimally at 4 of 6 HLA-A and B (at intermediate resolution by molecular typing) and DRB1 (at high resolution by molecular typing) loci with the patient, and HLA-matched at 3 of 6 HLA- A, B, DRB1 loci with each other (using same resolution of HLA typing as indicated above). There is no limitation on maximum cell dose.
* Have a high risk or refractory malignancy, or non-malignant disorder amenable to stem cell transplantation therapy.
* Meet eligibility requirements for allogeneic transplant per institutional standard practices.
* Have given written informed consent according to FDA guidelines (or consent of parent/legal guardian as applicable).
* Be <65 years of age at the time of study enrollment.

Exclusion Criteria:

* Have a consenting 8/8 or 10/10 allele matched, consenting, related or unrelated hematopoietic stem cell transplant (HSCT) donor.
* Have a life expectancy of less than 3 months.
* Have uncontrolled infections at time of cytoreduction.

Max Age: 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States